CLINICAL TRIAL: NCT03398590
Title: Promoting Lifestyle Changes With Mobile Health Technologies for Overweight or Obese Adults With Type 2 Diabetes - Feasibility and Acceptability Study
Brief Title: mHealth Intervention for Older Adults
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Boston College (Other)
Collaborators: Joslin Diabetes Center (Other)
Responsible Party: Principal Investigator, Yaguang Zheng, Assistant Professor, Boston College
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 17.192.01
Record Dates: First submitted 2017-10-31; First posted 2018-01-12 (Actual); Last update posted 2018-10-22 (Actual); Status verified 2018-10

CONDITIONS: Type2 Diabetes; Obesity
Keywords: Type 2 Diabetes; Obesity
MeSH Terms: conditions — Obesity; Diabetes Mellitus, Type 2

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- mHealth Intervention for Older Adults (Experimental): Pilot study to test the feasibility and acceptability of a self-regulation theory-based mHealth behavior intervention for overweight or obese older adults with T2DM.
  This is a one Group Pretest-Posttest Designed study. Ten participants will be recruited from Joslin Diabetes Center, Boston, MA. They will receive a 2-month, self-regulation theory-based weight loss intervention (five 60-minute, biweekly group sessions) and will be provided with a technology toolkit for self-monitoring including an (1) iPhone Plus, (2) the Lose It! app for self-monitoring of dietary intake, (3) Fitbit for self-monitoring of physical activity, (4) Bluetooth-enabled scale for daily weight, and (5) Bluetooth-enabled blood glucose monitor for testing blood glucose levels.
  Interventions: Behavioral: self-regulation theory-based mHealth behavior intervention

INTERVENTIONS:
Behavioral: self-regulation theory-based mHealth behavior intervention — Participants will receive a self-regulation theory-based mHealth behavior intervention (5 biweekly group sessions, 60 minutes /session). An experienced Certified Diabetes Educator from the Joslin Diabetes Center and PI (Dr. Zheng) who has been trained using self-regulation for weight loss will co-facilitate group sessions. The intervention combines diet modification and increased physical activity with a weekly weight loss goal as well as focuses on improving participants' three typical self-regulation strategies - self-monitoring, self-evaluation and self-reinforcement. Intervention duration will last 2 months with subsequent 1-month follow.

SUMMARY:
This is a pilot study to test the feasibility and acceptability of a self-regulation theory-based mHealth behavior intervention for overweight or obese older adults with T2DM.

DETAILED DESCRIPTION:
This is a pilot study to test the feasibility and acceptability of a self-regulation theory-based mHealth behavior intervention for overweight or obese older adults with T2DM. The main purpose of the intervention is to increase participants' awareness of their behavior patterns and to self-regulate their daily lifestyle behaviors using the results of self-monitoring of weight and blood glucose. This is a One Group Pretest-Posttest Designed study. Ten participants will be recruited from Joslin Diabetes Center, Boston, MA. They will receive a 2-month, self-regulation theory-based weight loss intervention (five 60-minute, biweekly group sessions) and will be provided with a technology toolkit for self-monitoring including an (1) iPhone Plus, (2) the Lose It! app for self-monitoring of dietary intake, (3) Fitbit for self-monitoring of physical activity, (4) Bluetooth-enabled scale for daily weight, and (5) Bluetooth-enabled blood glucose monitor for testing blood glucose levels. There will be a 1-month follow-up after intervention. Assessments will occur at baseline and the end of follow-up. The individual interviews will be conducted with the participants to learn about their experience of technology use to self-manage their weight and diabetes at the end of study.

ELIGIBILITY:
Inclusion Criteria:

* >=65 years of age;
* BMI between 27-40kg/m2
* Availability of wireless Internet service at home;
* Stable body weight during the previous year (i.e., ±10 pounds) ;
* Not being enrolled in another weight loss program in the past six months;
* Diagnosed with type 2 diabetes for at least 2 years;
* Prescribed insulin or oral medications for at least 1 year;
* No changes in medications for at least 6 months before enrolling in the study;
* Use the LoseIt! app on their computer or smartphone for the 5-day practice period;
* Able to read, write and speak English.

Exclusion Criteria:

* Planning frequent travel, vacations or relocation in next 3 months;
* Current use of weight loss medication;
* Have a history of bariatric surgery;
* Have participated in diabetes education in the previous 12 months;
* Are unable to walk 2 blocks, or had an amputation of a lower limb, severe arthritis or other medical condition that prevents walking for exercise;
* Have severe complications of diabetes, including renal disease (albumin/creatinine >300 μg /mg), severe peripheral diabetic neuropathy, severe peripheral vascular disease, symptomatic autonomic neuropathy, history of myocardial infarction, congestive heart failure, or other severe cardiac disease or severe hypertension (systolic blood pressure greater than 160/90 mmHg);
* Have a diagnosis of a serious mental illness, e.g. schizophrenia, bipolar disorder, substance abuse, and/or eating disorders;
* Have severe visual, hearing or cognitive impairments (e.g., dementia, intellectual disability);
* Unable or unwilling to use the mHealth technology equipment (toolkit) for data collection;
* Do not speak, read and write English.

Min Age: 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Enrollment: 9 (Actual)
Dates: Start 2017-04-12 (Actual); Primary Completion 2018-05-30 (Actual); Study Completion 2018-05-30 (Actual)

PRIMARY OUTCOMES:
Acceptability | From baseline to the end of study (up to 3 months)
  Actual Use of Technology will be defined as binary (use vs. nonuse) for each day based on data-stamp information. Then we will calculate percent days of use over time.

SECONDARY OUTCOMES:
Percent weight change | From baseline to the end of study (up to 3 months)
  Percent weight changes over 3 months
Steps | From baseline to the end of study (up to 3 months)
  Steps changes over 3 months
Calorie intake | Mean steps over 3 months
  Calorie intake changes over 3 months

CONTACTS AND LOCATIONS:
Overall Officials: Yaguang Zheng, PhD, Principal Investigator — Boston College Connell School of Nursing
Locations (1):
- Joslin Diabetes Center, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: Undecided